CLINICAL TRIAL: NCT03000582
Title: Pharmacokinetic Assessment of Acute Ingestion of Different Forms of Creatine
Brief Title: Assessment of Different Forms of Creatine
Acronym: NB3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Nutrabolt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB2014-0362F
Record Dates: First submitted 2016-12-14; First posted 2016-12-22 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Dietary Modification
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Creatine monohydrate (Experimental): 5 gm creatine monohydrate, 1.5 gm dextrose
  Interventions: Dietary Supplement: Creatine monohydrate
- Creatine nitrate-1 (Active Comparator): 1 gm creatine monohydrate, 0.5 gm nitrate, 5 gm dextrose
  Interventions: Dietary Supplement: Creatine nitrate-1
- Creatine nitrate-2 (Active Comparator): 2 gm creatine monohydrate, 1 gm nitrate, 3.5 gm dextrose
  Interventions: Dietary Supplement: Creatine nitrate-2
- Placebo (Placebo Comparator): 6.5 gm dextrose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine monohydrate — Creatine monohydrate (5.0 g creatine monohydrate, 1.5 g dextrose)
  Arms: Creatine monohydrate
Dietary Supplement: Creatine nitrate-1 — Creatine nitrate-1 (1.0 g creatine monohydrate, 0.5 g nitrate, 5.0 g dextrose)
  Arms: Creatine nitrate-1
Dietary Supplement: Creatine nitrate-2 — Creatine nitrate-2 (2.0 g creatine monohydrate, 1.0 g nitrate, 3.5 g dextrose)
  Arms: Creatine nitrate-2
Dietary Supplement: Placebo — Placebo (6.5 g dextrose)
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the pharmacokinetics of creatine nitrate supplementation.

DETAILED DESCRIPTION:
Creatine nitrate contains several nutrients that may increase anaerobic exercise performance. Theoretically, dietary supplementation of creatine nitrate during resistance training can improve the quality of training leading to greater changes in strength, power and fat free mass. Endothelial function measured by flow-mediated dilation (FMD), a non-invasive vascular health parameter that can be measured via ultrasonography, is a predictor of cardiovascular disease risk which precedes traditional risk markers. Diet, physical activity and pharmaceutical interventions can all impact vascular function and health. The purpose of this study is to determine the acute vascular response of creatine nitrate supplementation on FMD by analyzing the pharmacokinetics of creatine nitrate supplementation.

ELIGIBILITY:
Inclusion Criteria:

* you are an apparently healthy and recreationally active male between the ages of 18 and 40;

Exclusion Criteria:

* you have a history of treatment for metabolic disease (i.e., diabetes), hypertension, hypotension, thyroid disease, arrhythmia and/or cardiovascular disease;
* you are currently using prescription medications;
* you have a history of smoking;
* you drink excessively (i.e., 12 drinks per week or more);
* you have a recent history of creatine supplementation within six weeks of the start of supplementation;

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Examine creatine vs. creatine nitrate supplementation by assessing body water | One day
Examine creatine vs. creatine nitrate supplementation by assessing body composition | One day
Examine creatine vs. creatine nitrate supplementation by assessing serum creatine levels | One day
Examine creatine vs. creatine nitrate supplementation by assessing serum nitrate levels | One day
Examine creatine vs. creatine nitrate supplementation by assessing serum nitrite levels | One day
Examine creatine vs. creatine nitrate supplementation by assessing flow-mediated dilation (FMD) via ultrasonography | One day

SECONDARY OUTCOMES:
Measure standard clinical chemistry panels in the blood to evaluate safety | One day
Measure side effects to evaluate safety utilizing a side effects questionnaire | One day
Measure heart rate to evaluate safety | One day
Measure blood pressure to evaluate safety | One day

IPD SHARING:
Plan to Share IPD: No